CLINICAL TRIAL: NCT01672788
Title: Bioequivalence of Empagliflozin/Metformin (850 mg) Fixed Dose Combination Tablets Compared to Single Tablets Administered Together in Healthy Male and Female Volunteers Under Fed Conditions (an Open-label, Randomised, Single-dose, Four-way Crossover Study)
Brief Title: Demonstration of Bioequivalence of Empagliflozin and Metformin Given in One Tablet Compared to the Intake of Single Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1276.7; 2012-002277-65 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Metformin

ARMS (4):
- Test 1 (Experimental): fixed dose combination tablet
  Interventions: Drug: Empagliflozin + Metformin
- Reference 1 (Active Comparator): empagliflozin tablets and metformin tablet
  Interventions: Drug: Empagliflozin; Drug: Metformin
- Test 2 (Experimental): fixed dose combination tablet
  Interventions: Drug: Empagliflozin + Metformin
- Reference 2 (Active Comparator): empagliflozin tablet and metformin tablet
  Interventions: Drug: Metformin; Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — empagliflozin tablets and metformin tablet
  Arms: Reference 1
Drug: Empagliflozin + Metformin — fixed dose combination tablet (low)
  Arms: Test 2
Drug: Metformin — empagliflozin tablets and metformin tablet
  Arms: Reference 1
Drug: Metformin — empagliflozin tablet and metformin tablet
  Arms: Reference 2
Drug: Empagliflozin + Metformin — fixed dose combination tablet (low)
  Arms: Test 1
Drug: Empagliflozin — empagliflozin tablet and metformin tablet
  Arms: Reference 2

SUMMARY:
The primary objective of this trial is to establish bioequivalence of two FDC tablets and the single tablets when administered together after a high fat high caloric meal.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1276.7.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, randomized, 4-way crossover trial. 36 patients were randomised to one of 4 treatment sequences and treated. Each treatment period consisted of a single dose of medication followed by 72 hours of pharmacokinetic sampling, with a washout of at least 7 days between treatment periods.
Groups:
- T1 / R1 / T2 / R2: Patients received the 4 treatments in the following order:
  * Empa 12.5mg Fixed-dose: Fixed-dose tablet of 12.5mg empagliflozin plus 850mg metformin (T1)
  * Empa 12.5mg Free Dose: Free dose combination of 12.5mg empagliflozin (consisting of 1 tablet of 10mg and another of 2.5mg) and 850mg metformin (1 tablet) (R1)
  * Empa 5mg Fixed-dose: Fixed-dose tablet of 5mg empagliflozin plus 850mg metformin (T2)
  * Empa 5mg Free Dose: Free dose combination of 5mg empagliflozin (1 tablet) and 850mg metformin (1 tablet) (R2)
- R1 / T1 / R2 / T2: Patients received the 4 treatments in the following order:
  * Empa 12.5mg Free Dose: Free dose combination of 12.5mg empagliflozin (consisting of 1 tablet of 10mg and another of 2.5mg) and 850mg metformin (1 tablet) (R1)
  * Empa 12.5mg Fixed-dose: Fixed-dose tablet of 12.5mg empagliflozin plus 850mg metformin (T1)
  * Empa 5mg Free Dose: Free dose combination of 5mg empagliflozin (1 tablet) and 850mg metformin (1 tablet) (R2)
  * Empa 5mg Fixed-dose: Fixed-dose tablet of 5mg empagliflozin plus 850mg metformin (T2)
- T2 / R2 / T1 / R1: Patients received the 4 treatments in the following order:
  * Empa 5mg Fixed-dose: Fixed-dose tablet of 5mg empagliflozin plus 850mg metformin (T2)
  * Empa 5mg Free Dose: Free dose combination of 5mg empagliflozin (1 tablet) and 850mg metformin (1 tablet) (R2)
  * Empa 12.5mg Fixed-dose: Fixed-dose tablet of 12.5mg empagliflozin plus 850mg metformin (T1)
  * Empa 12.5mg Free Dose: Free dose combination of 12.5mg empagliflozin (consisting of 1 tablet of 10mg and another of 2.5mg) and 850mg metformin (1 tablet) (R1)
- R2 / T2 / R1 / T1: Patients received the 4 treatments in the following order:
  * Empa 5mg Free Dose: Free dose combination of 5mg empagliflozin (1 tablet) and 850mg metformin (1 tablet) (R2)
  * Empa 5mg Fixed-dose: Fixed-dose tablet of 5mg empagliflozin plus 850mg metformin (T2)
  * Empa 12.5mg Free Dose: Free dose combination of 12.5mg empagliflozin (consisting of 1 tablet of 10mg and another of 2.5mg) and 850mg metformin (1 tablet) (R1)
  * Empa 12.5mg Fixed-dose: Fixed-dose tablet of 12.5mg empagliflozin plus 850mg metformin (T1)
Period: Treatment Period 1 (3 Days)
Arm/Group | T1 / R1 / T2 / R2 | R1 / T1 / R2 / T2 | T2 / R2 / T1 / R1 | R2 / T2 / R1 / T1
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | T1 / R1 / T2 / R2 | R1 / T1 / R2 / T2 | T2 / R2 / T1 / R1 | R2 / T2 / R1 / T1
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (3 Days)
Arm/Group | T1 / R1 / T2 / R2 | R1 / T1 / R2 / T2 | T2 / R2 / T1 / R1 | R2 / T2 / R1 / T1
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | T1 / R1 / T2 / R2 | R1 / T1 / R2 / T2 | T2 / R2 / T1 / R1 | R2 / T2 / R1 / T1
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Treatment Period 3 (3 Days)
Arm/Group | T1 / R1 / T2 / R2 | R1 / T1 / R2 / T2 | T2 / R2 / T1 / R1 | R2 / T2 / R1 / T1
Started | 9 | 9 | 9 | 8
Completed | 9 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3 (7 Days)
Arm/Group | T1 / R1 / T2 / R2 | R1 / T1 / R2 / T2 | T2 / R2 / T1 / R1 | R2 / T2 / R1 / T1
Started | 9 | 9 | 9 | 8
Completed | 9 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 4 (3 Days)
Arm/Group | T1 / R1 / T2 / R2 | R1 / T1 / R2 / T2 | T2 / R2 / T1 / R1 | R2 / T2 / R1 / T1
Started | 9 | 9 | 9 | 8
Completed | 9 | 9 | 9 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total number of patients randomised and treated in the study. This was an open-label, randomized, 4-way crossover trial. 36 patients were randomised to one of 4 treatment sequences and treated. Each treatment period consisted of a single dose of medication followed by 72hours of pharmacokinetic sampling, with a washout of at least 7 days between treatment periods.
Arm/Group | Overall Study
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Empa: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity.
  In this endpoint, the "Measured values" shows inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40min, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration
Population: Pharmacokinetic (PK) set: All subjects who took at least 1 dose of investigational treatment, provided at least 1 observation for at least 1 primary PK endpoint, did not have important protocol violations relevant to the evaluation of relative bioavailability, did not vomit at or before 2 times median tmax and did not use restricted medications
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa 12.5mg Fixed-dose: Fixed-dose tablet of 12.5mg empagliflozin plus 850mg metformin
- Empa 12.5mg Free Dose: Free dose combination of 12.5mg empagliflozin (consisting of 1 tablet of 10mg and another of 2.5mg) and 850mg metformin (1 tablet)
- Empa 5mg Fixed-dose: Fixed-dose tablet of 5mg empagliflozin plus 850mg metformin
- Empa 5mg Free Dose: Free dose combination of 5mg empagliflozin (1 tablet) and 850mg metformin (1 tablet)
Arm/Group | Empa 12.5mg Fixed-dose | Empa 12.5mg Free Dose | Empa 5mg Fixed-dose | Empa 5mg Free Dose
Number analyzed (Participants) | 34 | 34 | 35 | 33
nmol*h/L | 2560 (25.5) | 2530 (29.5) | 986 (26.9) | 968 (23.9)
Statistical Analysis 1: Comparison: Empa 12.5mg Fixed-dose vs Empa 12.5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 12.5mg fixed-dose divided by empa 12.5mg free dose; ANOVA; Based on an ANOVA including the random effect subjects within sequences and the fixed effects sequence, period and treatment; Geometric Mean Ratio = 101.31, 90% CI 2-sided [96.89 to 105.93], Standard Deviation 10.7 — Standard deviation is actually the geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: Empa 5mg Fixed-dose vs Empa 5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 5mg fixed-dose divided by empa 5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 100.30, 90% CI 2-sided [97.40 to 103.29], Standard Deviation 7.0 — Standard deviation is actually the geometric coefficient of variation (gCV)

2. Primary Outcome: Metformin: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Empa 12.5mg Fixed-dose | Empa 12.5mg Free Dose | Empa 5mg Fixed-dose | Empa 5mg Free Dose
Number analyzed (Participants) | 34 | 34 | 35 | 33
ng*h/mL | 8640 (18.0) | 8450 (24.4) | 8520 (23.8) | 8560 (25.8)
Statistical Analysis 1: Comparison: Empa 12.5mg Fixed-dose vs Empa 12.5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 12.5mg fixed-dose divided by empa 12.5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 101.61, 90% CI 2-sided [97.94 to 105.41], Standard Deviation 8.8 — Standard deviation is actually the gCV
Statistical Analysis 2: Comparison: Empa 5mg Fixed-dose vs Empa 5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 5mg fixed-dose divided by empa 5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 98.56, 90% CI 2-sided [94.24 to 103.08], Standard Deviation 10.8 — Standard deviation is actually the gCV

3. Secondary Outcome: Empa: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point.
  In this endpoint, the "Measured values" shows inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa 12.5mg Fixed-dose | Empa 12.5mg Free Dose | Empa 5mg Fixed-dose | Empa 5mg Free Dose
Number analyzed (Participants) | 34 | 34 | 35 | 33
nmol*h/L | 2520 (25.1) | 2490 (29.3) | 963 (27.1) | 946 (24.2)
Statistical Analysis 1: Comparison: Empa 12.5mg Fixed-dose vs Empa 12.5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 12.5mg fixed-dose divided by empa 12.5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 101.20, 90% CI 2-sided [96.89 to 105.71], Standard Deviation 10.4 — Standard deviation is actually the geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: Empa 5mg Fixed-dose vs Empa 5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 5mg fixed-dose divided by empa 5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 100.31, 90% CI 2-sided [97.41 to 103.30], Standard Deviation 7.0 — Standard deviation is actually the gCV

4. Primary Outcome: Empa: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of the analyte in plasma, per period.
  In this endpoint, the "Measured values" shows inter-individual variabilities, whereas the statistical analyses show intra-individual variabilities.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa 12.5mg Fixed-dose | Empa 12.5mg Free Dose | Empa 5mg Fixed-dose | Empa 5mg Free Dose
Number analyzed (Participants) | 34 | 34 | 35 | 33
nmol/L | 266 (20.3) | 258 (21.3) | 103 (22.1) | 101 (24.4)
Statistical Analysis 1: Comparison: Empa 12.5mg Fixed-dose vs Empa 12.5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 12.5mg fixed-dose divided by empa 12.5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 102.70, 90% CI 2-sided [98.75 to 106.81], Standard Deviation 9.4 — Standard deviation is actually the geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: Empa 5mg Fixed-dose vs Empa 5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 5mg fixed-dose divided by empa 5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 100.97, 90% CI 2-sided [95.94 to 106.27], Standard Deviation 12.3 — Standard deviation is actually the gCV

5. Primary Outcome: Metformin: Maximum Measured Concentration (Cmax)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Empa 12.5mg Fixed-dose | Empa 12.5mg Free Dose | Empa 5mg Fixed-dose | Empa 5mg Free Dose
Number analyzed (Participants) | 34 | 34 | 35 | 33
ng/mL | 1080 (16.4) | 1080 (19.6) | 1090 (16.5) | 1100 (17.5)
Statistical Analysis 1: Comparison: Empa 12.5mg Fixed-dose vs Empa 12.5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 12.5mg fixed-dose divided by empa 12.5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 99.64, 90% CI 2-sided [95.39 to 104.09], Standard Deviation 10.5 — Standard deviation is actually the geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: Empa 5mg Fixed-dose vs Empa 5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 5mg fixed-dose divided by empa 5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 97.89, 90% CI 2-sided [93.82 to 102.15], Standard Deviation 10.2 — Standard deviation is actually the gCV

6. Secondary Outcome: Metformin: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Empa 12.5mg Fixed-dose | Empa 12.5mg Free Dose | Empa 5mg Fixed-dose | Empa 5mg Free Dose
Number analyzed (Participants) | 34 | 34 | 35 | 33
ng*h/mL | 8370 (18.1) | 8190 (24.1) | 8280 (23.2) | 8320 (25.2)
Statistical Analysis 1: Comparison: Empa 12.5mg Fixed-dose vs Empa 12.5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 12.5mg fixed-dose divided by empa 12.5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 101.51, 90% CI 2-sided [97.95 to 105.21], Standard Deviation 8.6 — Standard deviation is actually the geometric coefficient of variation (gCV)
Statistical Analysis 2: Comparison: Empa 5mg Fixed-dose vs Empa 5mg Free Dose; Test type: Non-Inferiority or Equivalence — Considered characteristic is empa 5mg fixed-dose divided by empa 5mg free dose; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 98.57, 90% CI 2-sided [94.50 to 102.81], Standard Deviation 10.1 — Standard deviation is actually the gCV

ADVERSE EVENTS:
Time Frame: Treatment period and following washout period, up to 35 days
Arm/Group | Empa 12.5mg Fixed-dose | Empa 12.5mg Free Dose | Empa 5mg Fixed-dose | Empa 5mg Free Dose
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 14/35 | 13/36 | 14/34 | 9/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa 12.5mg Fixed-dose (N=35) | Empa 12.5mg Free Dose (N=36) | Empa 5mg Fixed-dose (N=34) | Empa 5mg Free Dose (N=35)
Diarrhoea (Gastrointestinal disorders) | 8 | 8 | 5 | 7
Nausea (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Nasopharyngitis (Gastrointestinal disorders) | 3 | 2 | 4 | 0
Headache (Nervous system disorders) | 5 | 3 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.